CLINICAL TRIAL: NCT07348575
Title: A Multicenter, Prospective, Randomized, Controlled Study of Decitabine in Combination With R-CHOP for Initial Treatment of EBV+ Diffuse Large B-cell Lymphoma
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR/AF/SG-05/1.1
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-01

CONDITIONS: Lymphoma, Large-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — R-CHOP protocol; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decitabine in combination with R-CHOP (Experimental): Decitabine in combination with R-CHOP
  Interventions: Drug: Decitabine in combination with R-CHOP
- R-CHOP (Active Comparator): R-CHOP
  Interventions: Drug: R-CHOP

INTERVENTIONS:
Drug: R-CHOP — Decitabine in combination with R-CHOP
  Arms: R-CHOP
Drug: Decitabine in combination with R-CHOP — Decitabine in combination with R-CHOP
  Arms: Decitabine in combination with R-CHOP

SUMMARY:
This trial was a prospective, multicenter, randomized, controlled Phase III clinical design to compare the efficacy and safety of decitabine combined with R-CHOP (R-CHOP-D) versus R-CHOP in the treatment of primary EBV+ diffuse large B-cell lymphoma (DLBCL).

Sixty patients were randomized 1:1 into R-CHOP-D (trial group) or R-CHOP (control group). The trial consisted of a screening period (days -28 to -1), a treatment period, and a follow-up period (2 years after the end of the last trial).

ELIGIBILITY:
Inclusion Criteria:

1. Initial treatment of diffuse large B-cell lymphoma (DLBCL) confirmed by tumor histopathology with at least one lesion on either axis More than 1.5 cm, sufficient specimens for second-generation sequencing or single-cell sequencing;
2. Age > 18 years old, < 80 years old, gender unlimited;
3. EBER+ or peripheral blood EBV-DNA of pathological specimen was greater than 103copy/ml;
4. Patients judged by the investigator to have a life expectancy of at least 6 months;
5. The patient or his legal representative must provide written informed consent prior to any research special examination or procedure.
6. Signed written informed consent before screening.

Exclusion Criteria:

1. Have previously received systemic or local treatment including chemotherapy;
2. Previously received autologous stem cell transplantation;
3. Previous history of other malignant tumors, except skin basal cell carcinoma and cervical carcinoma in situ;
4. Accompanied by uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, connective tissue diseases and serious infectious diseases;
5. Lymphoma involves the central nervous system;
6. Primary mediastinal large B-cell lymphoma;
7. Left ventricular ejection fraction < 50%;
8. Laboratory test values at the time of screening: (unless due to lymphoma);

   1. Neutrophils < 1.5 x 109/L;
   2. Platelet < 75 x 109/L;
   3. ALT or AST were 2 times higher than the upper limit of normal, AKP and bilirubin were 1.5 times higher than the upper limit of normal;
   4. creatinine levels higher than 1.5 times the upper limit of normal;
9. Patients with mental illness or other patients known or suspected to be unable to fully comply with the study protocol;
10. Pregnant or lactating women;
11. Known human immunodeficiency virus (HIV) infection, or active hepatitis B or C virus infection (polymerase chain Reaction [PCR] showed positive results). If the HbsAg test result is positive, HBV DNA test should be performed, if the HBV DNA<103IU/ml, can be enrolled. If HBsAg test results are negative, but HBcAb test is positive (regardless of HBsAb status), HBV DNA test is also required, and HBV DNA<103 IU/ml can be enrolled. If the patient's HCV antibody is positive, the HCV RNA is detected by PCR. If positive, the exclusion criteria are met.
12. Other concurrent and uncontrolled medical conditions that the investigator believes will affect the patient's participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided